CLINICAL TRIAL: NCT05219357
Title: Ayurveda Based Intervention for Patients in Acute Psychiatric Crisis: Pilot Trial Using Community-Based Participatory Research
Brief Title: Ayurveda Based Intervention for Patients in Acute Psychiatric Crisis Situations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarogyam UK (Other)
Collaborators: NMP Medical Research Institute (Other); Croydon Ayurveda Centre (Unknown); Active Naturals Limited (Unknown); AVP Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP1873-92
Record Dates: First submitted 2022-01-06; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Psychiatric Disorder
Keywords: Ayurveda; Mental Health; Emergencies; Community Based Participatory Research
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Emergencies | interventions — Medicine, Ayurvedic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (UCG) (Active Comparator): The usual care control group received care only on hospital wards during episodes
  Interventions: Drug: Usual-Care
- Ayu Care Group (ACG) (Other): Multidisciplinary Ayurveda based treatment team aimed to manage acute crises of patients in the community settings or at their home if feasible.
  Interventions: Other: Ayu-Care

INTERVENTIONS:
Other: Ayu-Care — Ayurveda treatment modalities includes three parts to manage mental health Satwawajay Chikitsa, Yuktivyapashray and Daivyapashray Chikitsa. It is based on personalised whole person approach.
  Other Names: Ayurveda
  Arms: Ayu Care Group (ACG)
Drug: Usual-Care — Management strategies includes restraints, emergency medications, behavioral interventions, with a special focus on the pharmacological interventions.
  Arms: Usual Care Group (UCG)

SUMMARY:
For patients undergoing a psychiatric crisis, hospitalisation is required. In developing countries specially in sub-urban or rural areas, most patients don't access intensive care. In India, AYUSH system of medical care is widely used, including crisis resolution and community treatment have been widely implemented in various mental health systems. However, evidence to support their effectiveness has remained very low.

Present study is designed as community based participatory research, where Ayurveda treatment , a short-term, specialised, crisis intervention is provided by community outreach team.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with a psychiatric complaint.
* Male or female patients at least 18 years of age.
* Each patient, or a patient's legal representative (as allowed by local law), must understand the nature of the study and must agree to study enrollment.

Exclusion Criteria:

* Patients who have delirium or dementia
* Prisoners
* Pediatric patients
* Elderly patients
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Brief Symptom Inventory | Change from baseline to 48 hours and 7th-days of intervention
  Brief Symptom Inventory was used to assess self-report of psychological problems and symptom severity
Length of Emergency hospital stay | Hours spent in the Emergency Department (ED), measured at the index ED visit (Day 0)
  Length of stay is defined as the time between patient triage and discharge from the emergency department

SECONDARY OUTCOMES:
The Kessler Psychological Distress Scale (K10) | Change from baseline to 3rd and 7th-days of intervention
  The K10 comprises 10 items that rate symptoms along the anxiety-depression spectrum, with a five point Likert response, where one is 'none of the time' to five 'all of the time.
The Psychological Outcome Profiles instrument | From Baseline to 3rd and 7th-days of intervention
  To measure participant-generated outcomes comprising four items on 6 scale (0-5) 0 = not at all affected' to '5 = severely affected.
Agitation Calmness Evaluation Scale (ACES) | From Baseline to 48 hours and 7th-days of intervention
  The ACES consists of a single item that rates overall agitation at the time of patients observations on 9 scale (1=marked agitation, 4=normal behaviour, 9= unarousable)
Positive and Negative Syndrome Scale; | From Baseline to 48 hours and 7th-days of intervention
  The tool consists of 5 items: excitement, tension, hostility, being uncooperative, and poor impulse control. Each item is scored on 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme)
Satisfaction with acute care | From Baseline to 3rd and 7th-days of intervention
  Measured on 5-point scale, completed by the participant using the Service Satisfaction Scale 10 (SSS-10), from 1 (No, definitely not) to five (Yes, definitely)
Side effects | From Index ED visit to 30 days
  The frequency of any side effects or adverse events experienced by individuals to both intervention group on 4 point scale (landing from absent=0 to severe=3)
Medication use | From Index ED visit to 30 days
  Daily doses and classes of medications (e.g. antipsychotics, mood stabilizers, benzodiazepines, etc.) or other treatments or interventions prescribed per individual

OTHER OUTCOMES:
Death by Suicide | From Index ED visit to 30 days
  Death by suicide within 30 days of the index ED visit

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Study Director — Aarogyam (UK) CIC; Venkata N Joshi, Study Chair — Croydon Ayurveda Centre; Maël Voegeli, Principal Investigator — AVP Research Foundation; Skanthesh Lakshmanan, Study Chair — NMP Medical Research Institute
Locations (2):
- India (2):
  - Gyansanjeevani, Jaipur, Rajasthan
  - NMP Medical Research Institite, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No
Individual Participants Data will not be available to other researchers. Data will only be shared through publications and presentations on study completion.